CLINICAL TRIAL: NCT02044835
Title: The Evaluation Studies of Curative Effect of Fu-zheng-qu-zhuo Oral Liquid in Treatment of Ischemic Nephropathy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: lishen58173
Record Dates: First submitted 2014-01-22; First posted 2014-01-24 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Atherosclerotic Renal Artery Stenosis
Keywords: atherosclerotic renal artery stenosis, herbal medicine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OMT controll (Placebo Comparator): placebo 20 ml every time, three times a day, combined with optimal medical therapy of internal medicine, including anti-platelet therapy and other protocol-driven medical therapies to control blood pressure and glucose and lipid levels in accordance with guidelines.
- herbal treatment (Experimental): Fu-zheng-qu-zhuo oral liquid ( herbal medicine) 20 ml every time, three times a day,combined with optimal medical therapy of internal medicine, including anti-platelet therapy and other protocol-driven medical therapies to control blood pressure and glucose and lipid levels in accordance with guidelines.
  Interventions: Drug: Fu-zheng-qu-zhuo oral liquid

INTERVENTIONS:
Drug: Fu-zheng-qu-zhuo oral liquid — Fu-zheng-qu-zhuo oral liquid was composed of Ginseng, Astragalus, Angelica root, Tuckahoe, Rhubarb, etc. It was producted by manufacturing laboratory of Guang'anmen Hospital, China Academy of Chinese Medical Science (License code: 京药制字Z20063242)
  Arms: herbal treatment

SUMMARY:
• Background: Since evidence show that renal-artery stenting did not confer a significant benefit with respect to the prevention of clinical events when added to comprehensive, multifactorial medical therapy in people with atherosclerotic renal-artery stenosis[1], the aim of our study was to confirm Fu-zheng-qu-zhuo (FZQZc) oral liquid, a herbal medicine, combined with optimal medical therapy of internal medicine (OMT), including anti-platelet therapy and other protocol-driven medical therapies to control blood pressure and glucose and lipid levels in accordance with guidelines,resulted in greater renal function protection in patients with atherosclerotic renal artery stenosis ( ARAS) compared with OMT alone.

Methods : A randomized, placebo-controlled, single centre clinical design. Sixty patients with diagnosed atherosclerotic renal artery stenosis and had chronic kidney disease stage 3 will be recruited, and will be randomized into two groups in a 1:1 ratio ( FZQZ and placebo Group, 30 respectively). FZQZ Oral liquid or placebo 20 ml every time, three times a day for different groups, meanwhile, all participants in both treatment groups received OMT, 6 months therapeutic period. Serum creatinine, estimated glomerular filtration rate(eGFR), urine protein, and cardiovascular and renal events (a composite end point of death from cardiovascular or renal causes, myocardial infarction, stroke, hospitalization for congestive heart failure, progressive renal insufficiency, or the need for renal-replacement therapy) will be compared between the Groups as the outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Met the ARAS diagnosis: renal angiography or magnetic resonance angiography (MRA) shows renal artery with unilateral or bilateral stenosis at least 50%，and with artery atheromatous plague;
2. Meeting with the diagnostic criteria of the K/DOQI chronic kidney disease （eGFR<90ml/min）：light or moderate damage to kidney function，Scr<265.2µmol/L(3.0mg/dl).

Exclusion Criteria:

1. Patients with renal artery stenosis which had been suspected or final diagnosed to be Fibromuscular dysplasia or Takayasu arteritis;
2. Blood pressure did not meet the target (<140/90mmHg) after combinedly taking more three kinds of antihypertensive agents with maximum dose;
3. Poor control of blood sugar in patients with Diabetes ( glycosylated hemoglobin 8.0% or higher in the recent month);
4. History of peptic ulcer，with Gastrointestinal bleeding in the recent 6 months;
5. decompensated cirrhosis;
6. Hematologic disease or bleeding tendency;
7. Repeated episodes of pulmonary edema, congestive heart failure, acute myocardial infarction, cerebral infarction and cerebral hemorrhage in recent 3 months;
8. Suffering from malignant tumor and predicting life span less than 1 year.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
estimated glomerular filtration rate filtration rate | six month
  the change of eGFR during the observation period

SECONDARY OUTCOMES:
cardiovascular and renal events (a composite end point of death from cardiovascular or renal causes( myocardial infarction, stroke, hospitalization for congestive heart failure, progressive renal insufficiency, or the need for renal-replacement therapy) | six month

OTHER OUTCOMES:
urine protein | six month

CONTACTS AND LOCATIONS:
Locations (1):
- Guang anmen Hospital,China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China